CLINICAL TRIAL: NCT04304274
Title: Early and Late Postoperative Analgesia and Recovery Effects of Programmed Intermittent Bolus Infusion of Thoracic Paravertebral Block for Hepatectomy: A Prospective, Randomized, Double-blinded, Controlled Study
Brief Title: Programmed Intermittent Bolus Infusion of Thoracic Paravertebral Block for Hepatectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cui Xulei (Other)
Responsible Party: Sponsor-Investigator, Cui Xulei, Professor, Peking Union Medical College Hospital
Organization: Peking Union Medical College Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: PTPVB-H
Record Dates: First submitted 2020-03-05; First posted 2020-03-11 (Actual); Last update posted 2022-02-18 (Actual); Status verified 2022-02

CONDITIONS: Paravertebral Block; Hepatectomy; Analgesia; Postoperative Recovery
MeSH Terms: conditions — Agnosia | interventions — Control Groups; Analgesia, Patient-Controlled; Morphine

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PTPVB-ropivacaine (Experimental): Programmed intermittent bolus infusion of a thoracic paravertebral block with ropivacaine and patient-controlled analgesia with morphine
  Interventions: Procedure: Paravertebral block-ropivacaine; Drug: patient controlled analgesia with morphine
- PTPVB-saline (Placebo Comparator): Programmed intermittent bolus infusion of a thoracic paravertebral block with saline and patient-controlled analgesia with morphine
  Interventions: Procedure: Paravertebral block-saline; Drug: patient controlled analgesia with morphine

INTERVENTIONS:
Procedure: Paravertebral block-ropivacaine — Inject 25 ml 0.5% ropivacaine in the T8 paravertebral space followed with catheter insertion and continuous 0.2% ropivacaine infusion(infusion rate: 0.125ml/kg/pulse,1pulse/h)
  Other Names: PVB group
  Arms: PTPVB-ropivacaine
Procedure: Paravertebral block-saline — Inject 25 ml 0.9% saline in the T8 paravertebral space followed with catheter insertion and continuous 0.9% saline infusion(infusion rate: 0.125ml/kg/pulse,1pulse/h)
  Other Names: Control group
  Arms: PTPVB-saline
Drug: patient controlled analgesia with morphine — Morphine was given as intravenous patient-controlled analgesia bolus: 1-2mg, lock time: 5min, 1h limitation: 8mg
  Other Names: PCIA

SUMMARY:
Hepatectomy induces moderate to severe postoperative pain. Patient-controlled intravenous analgesia has been used in many medical centers for post-hepatectomy analgesia, but the effects are limited and often cause undesirable adverse effects.

Regional Block has been used for postoperative analgesia in many surgeries. Some studies suggest that regional analgesia has an opioid-sparing effect and can reduce the incidence of chronic pain. Also, the programmed intermittent bolus infusion is better than continuous infusion, with less analgesic consumption and fewer adverse effects.

Studies on the early and late postoperative analgesia and recovery effects of paravertebral block for open hepatectomy are scarce. Therefore, the investigators aim to conduct a prospective, randomized, subject and assessor-blinded, parallel-group, placebo-controlled study to test the hypothesis that the programmed intermittent bolus infusion of right thoracic paravertebral block reduces postoperative intravenous analgesic use and pain scores and improved patients' satisfaction.

DETAILED DESCRIPTION:
This study aims to compare the early postoperative morphine consumptions, pain scores, rescue analgesics, adverse effects and recovery indices, and the late postoperative life quality between patients with and without paravertebral block.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-70 yrs
* American Society of Anesthesiologists physical statusⅠ-Ⅲ
* Undergo hepatectomy with J-shape subcostal incision
* Informed consent

Exclusion Criteria:

* A known allergy to the drugs being used
* Coagulopathy, on anticoagulants
* Analgesics intake, history of substance abuse
* Participating in the investigation of another experimental agent
* Unable to cooperate, eg. inability to properly describe postoperative pain to investigators

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2020-03-10 (Actual); Primary Completion 2021-06-10 (Actual); Study Completion 2021-12-10 (Actual)

PRIMARY OUTCOMES:
Postoperative 48hrs morphine | Postoperative 48 hours
  Cumulate morphine consumption 48 hours after hepatectomy

SECONDARY OUTCOMES:
Heart rate | During the operation
  The average value of the heart rate during the operation measured at 10 minutes interval
Mean blood pressure | During the operation
  The average value of the mean blood pressure (=1/3 systolic pressure + 2/3 diastolic pressure) during the operation measured at 10 minutes interval.
Sevoflurane concentration | During the operation
  The average value of the sevoflurane concentration during the operation measured at 10 minutes interval
Intraoperative medication dose | During the operation
  Doses of fentanyl, ephedrine, atrophin, phylepherine and urapidil used during the operation
Fluid volumes | During the operation
  Fluid volumes including volumes of crystalloid, colloid, red blood cells, plasma, platelet, Urine and hemorrhage.
Awake and extubation time | At the end of the operation
  Time from stop of sevoflurane use to patient awake and extubation.
Postoperative morphine consumption | Postoperative 2, 4, 12, 24hours
  Cumulative morphine consumption at 2, 4, 12, 24 hours after hepatectomy
Operation time | During the operation
  Time from the start to the end of the operation
The pain scores(at rest and with cough) determined by the numeric rating scale | Postoperative 0, 2, 4, 12, 24 and 48 hours
  NRS is an internationally recognized pain scale with 11 points ranging from 0 to 10 points, with 0 defined as no pain and 10 defined as the worst pain imaginable.
Adverse effects | Postoperative 0-48 hours
  Adverse effects of morphine including nausea, vomiting, pruritus and respiratory depression, bowel movement and Foley catheter removal.
Rescue analgesia | Postoperative 0-48hours
  Times of rescue analgesia
Postoperative recovery indices | Postoperative 48 hours
  Postoperative recovery indices including drowsiness, thirsty, cold feeling, cognitive decline and shiver evaluated using a 0-3 points Likert scale, with 0 defined as none, 1 defined as mild, 2 defined as moderate and 3 defined as severe.
Satisfaction indices | Postoperative 48 hours
  Emergence, analgesia and overall satisfaction evaluated using a 1-5 points Likert scale, with 1 defined as very unsatisfied, 2 defined as unsatisfied, 3 defined as no comments, 4 defined as satisfied and 5 defined as very satisfied.
Length of hospital stay | Two weeks after hospital discharge
  Number of in-hospital days from admission to discharge
Chronic recovery data | Postoperative 3 months
  Chronic recovery data including incidence of pain, numbness, hypoesthesia and sleep disorder
Chronic pain characteristics | Postoperative 3 months
  Incidence of difference types of pain including throbbing, aching, pricking and stabbing.
Chronic pain NRS score | Postoperative 3 months
  NRS is an internationally recognised pain scale with 11 points ranging from 0 to 10 points, with 0 defined as no pain and 10 defined as the worst pain imaginable.

CONTACTS AND LOCATIONS:
Overall Officials: Xulei Cui, MD, Principal Investigator — Peking Union Medical College Hospital
Locations (1):
- Peking Union Medical College Hospital, Beijing, China

REFERENCES:
- [Derived] Wang J, Cui X, Zhang Y, Sang X, Shen L. The effects of intermittent bolus paravertebral block on analgesia and recovery in open hepatectomy: a randomized, double-blinded, controlled study. BMC Surg. 2023 Aug 5;23(1):218. doi: 10.1186/s12893-023-02125-0. PMID 37543575